CLINICAL TRIAL: NCT00322595
Title: An International, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Active-Controlled Study of the Efficacy and Safety of Sustained-Release Quetiapine Fumarate (Seroquel SR™ ) in the Treatment of Generalized Anxiety Disorder (SILVER)
Brief Title: Efficacy and Safety Study of Seroquel SR in the Treatment of Generalized Anxiety Disorder
Acronym: SILVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00011; 2005-005054-46; Silver
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2007-12

CONDITIONS: Generalized Anxiety Disorder
Keywords: Anxiety; GAD
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Quetiapine Fumarate; Paroxetine

INTERVENTIONS:
Drug: Quetiapine fumarate
Drug: Paroxetine

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of (SEROQUEL SR™ ) quetiapine fumarate sustained-release (SR) compared to placebo in the treatment of anxiety symptoms in patients with generalized anxiety disorder (GAD).

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 65 years;
* A diagnosis of generalized anxiety disorder;
* Absence of current episode of major depression.

Exclusion Criteria:

* The presence or history of schizophrenia and other psychotic disorders;
* Hypertension;
* A current diagnosis of cancer, unless in remission for at least 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2006-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy compared to placebo in the treatment of anxiety symptoms in patients with generalized anxiety disorder (GAD) at Day 57 (= end of treatment).

SECONDARY OUTCOMES:
To evaluate efficacy by evaluating response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Seroquel Medical Science Director, Study Director — AstraZeneca
Locations (86):
- Argentina (7):
  - Research Site, City Bell, Buenos Aires
  - Research Site, Godoy Cruz, Mendoza Province
  - Research Site, Mendoza, Mendoza Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
- Bulgaria (6):
  - Research Site, Kardzhali
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vratsa
- Canada (15):
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Miramichi, New Brunswick
  - Research Site, Corner Brook, Newfoundland and Labrador
  - Research Site, Sydney, Nova Scotia
  - Research Site, Brantford, Ontario
  - Research Site, Chatham, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Orléans, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Czechia (7):
  - Research Site, Brno
  - Research Site, Litoměřice
  - Research Site, Olomouc
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Prerova
  - Research Site, Prostojov
- Denmark (3):
  - Research Site, Aarhus
  - Research Site, Copenhagen
  - Research Site, Frederiksberg
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Jarvenpaa
  - Research Site, Salo
  - Research Site, Turku
- France (9):
  - Research Site, Angoulême
  - Research Site, Arcachon
  - Research Site, Cherbourg
  - Research Site, Élancourt
  - Research Site, La Valette-du-Var
  - Research Site, Le Pecq
  - Research Site, Nîmes
  - Research Site, Rennes
  - Research Site, Toulouse
- Germany (7):
  - Research Site, Bad Saarow
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, München
  - Research Site, Siegen
- Mexico (3):
  - Research Site, Distrito Federal
  - Research Site, Guadalajara
  - Research Site, México
- Norway (3):
  - Research Site, Brattvåg
  - Research Site, Oslo
  - Research Site, Paradis
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Piteşti
  - Research Site, Sibiu
- Slovakia (6):
  - Research Site, Bojnice
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Košice
  - Research Site, Liptovský Mikuláš
  - Research Site, Zilina-Bytcica
- South Africa (4):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Pretoria
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Salamanca
- Sweden (5):
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Sundsvall
  - Research Site, Uppsala

REFERENCES:
- [Derived] Montgomery SA, Locklear JC, Svedsater H, Eriksson H. Efficacy of once-daily extended release quetiapine fumarate in patients with different levels of severity of generalized anxiety disorder. Int Clin Psychopharmacol. 2014 Sep;29(5):252-62. doi: 10.1097/YIC.0000000000000026. PMID 24394383
- [Derived] Stein DJ, Bandelow B, Merideth C, Olausson B, Szamosi J, Eriksson H. Efficacy and tolerability of extended release quetiapine fumarate (quetiapine XR) monotherapy in patients with generalised anxiety disorder: an analysis of pooled data from three 8-week placebo-controlled studies. Hum Psychopharmacol. 2011 Dec;26(8):614-28. doi: 10.1002/hup.1256. Epub 2011 Dec 6. PMID 22143997
- [Derived] Bandelow B, Chouinard G, Bobes J, Ahokas A, Eggens I, Liu S, Eriksson H. Extended-release quetiapine fumarate (quetiapine XR): a once-daily monotherapy effective in generalized anxiety disorder. Data from a randomized, double-blind, placebo- and active-controlled study. Int J Neuropsychopharmacol. 2010 Apr;13(3):305-20. doi: 10.1017/S1461145709990423. Epub 2009 Aug 20. PMID 19691907